CLINICAL TRIAL: NCT02805569
Title: Comparison of Intubation Conditions of the Articulating Stylet and Intubating Stylet Guided Videolaryngoscopy in Patients With Difficult Airway
Brief Title: Comparison of Intubation Conditions of the Articulating Stylet and Intubating Stylet Guided Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Associated profesor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 27/28
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Difficult Intubation
Keywords: videolaryngoscope; intubation stylet; articulating stylet; difficult airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): articulating stylet
  Interventions: Device: articulating stylet
- group C (Active Comparator): conventional stylet
  Interventions: Device: conventional stylet

INTERVENTIONS:
Device: articulating stylet — patient who intubated with articulating stylet
  Arms: Group A
Device: conventional stylet — patient who intubated with conventional stylet
  Arms: group C

SUMMARY:
Indirect videolaryngoscopes provide an improved view of the glottis. Unfortunately enhanced video blade angulation leads to difficulty in passage of the endotracheal tube (ETT) towards the larynx around the steep blade angulation despite adequate visualization of the glottis. Pre-shaping the ETT with the rigit malleable stylet is recommended. The investigators hypothesized that using articulating stylet (AS) would enhance first attempt intubation, shorten the intubation time, reduce the possibility of the soft tissue trauma compared to conventional intubation stylet (IS) in patients with difficult airway .

DETAILED DESCRIPTION:
Patients with known airway difficulty (anticipated difficult airway (ADA) score >6) will be included to the study.

All patients will receive general anesthesia for a variety of elective surgical procedure. Tracheal intubation will be performed by senior anesthesiologist. Patients will be intubated using AS-videolaryngoscope (n= 24) or IS-videolaryngoscope (n=24) randomly. Patients demographic details (age 18-65 yr, body mass index, ASA phisical status), ADA scores, Cormack-Lehane scores, intubation difficulty scores, intubation attempts, intubation time, hemodynamic variables, sore throat, anesthesiologists satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 physical status (Anticipated difficult airway) ADA scores >6 Elective surgery

Exclusion Criteria:

* ASA 3-4 physical status Immobilizedcervical spine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
intibation time | Through intubation completion, an avarage of 5 minutes
  Total intubation time (second)

SECONDARY OUTCOMES:
tracheal intubation attempts | Through intubation completion, an avarage of 5 minutes
  number of intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özkan, MD, Principal Investigator — Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Ankara, Turkey
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Ankara, Turkey, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Result] Suppan L, Tramer MR, Niquille M, Grosgurin O, Marti C. Alternative intubation techniques vs Macintosh laryngoscopy in patients with cervical spine immobilization: systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2016 Jan;116(1):27-36. doi: 10.1093/bja/aev205. Epub 2015 Jun 30. PMID 26133898